CLINICAL TRIAL: NCT05787847
Title: Financial Incentives to Promote Stimulant Abstinence in a Community-Based Syringe Exchange Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, richard rawson, Research Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVermont - FI for StimUD
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stimulant Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education (Other)
  Interventions: Behavioral: Health Education
- Health Education plus Incentives for Abstinence (Experimental)
  Interventions: Behavioral: Incentives for Abstinence; Behavioral: Health Education

INTERVENTIONS:
Behavioral: Incentives for Abstinence — Participants in the incentives for abstinence condition will have the opportunity to earn financial incentives for abstaining from stimulant use.
  Arms: Health Education plus Incentives for Abstinence
Behavioral: Health Education — The Health Education condition is based on a previous intervention used as a control in a number of other studies. Sessions consist of an educational program addressing a variety of health, wellness, and lifestyle topics adapted from a previously implemented wellness manual.

SUMMARY:
The goal of this randomized control pilot study is to learn about a financial incentives intervention among individuals who use stimulants and take part in a community-based syringe exchange program. The main question it aims to answer is how financial incentives for not using stimulants will impact stimulant use. Participants in the experimental group will have the opportunity to earn financial incentives for providing a negative urine sample for stimulants using a point-of-care test, which indicates abstinence from stimulant use, along with health education on the health risks of stimulant use and substance injection. Researchers will compare the experimental group to the control group who will receive health education on the health risks of stimulants use and injection.

DETAILED DESCRIPTION:
The investigators are proposing a two condition, parallel groups, randomized control pilot study to evaluate the efficacy of a financial incentives intervention among individuals who use stimulants and take part in a community-based syringe exchange program. The study design will include recruiting service recipients who already participate in programs offered by a syringe exchange program.The experimental group will have the opportunity to earn financial incentives contingent on providing a negative urine sample for stimulants using a point-of-care test, which indicates abstinence from stimulant use, in addition to health education on the health risks of stimulant use and substance injection. The control group will receive health education on the health risks of stimulants use and injection. All participants will participate in their syringe exchange services as usual. The investigators chose the health education as the control because participants across both conditions already receive the services provided by the syringe exchange program. Moreover, this control condition will help control for a potential type of between-groups variability.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older
* report using stimulants in the past 30 days
* meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis for stimulant use disorder at a moderate or severe level (i.e., 6 or more of the 11 criteria)
* participation in services at syringe exchange program

Exclusion Criteria:

* failure to meet one or more inclusionary criteria
* individuals who are cognitively impaired by their drug use or psychiatric conditions that could preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Howard Center, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Inclusion Criteria:
  * be 18 years or older
  * report using stimulants in the past 30 days
  * meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis for stimulant use disorder at a moderate or severe level
  * participation in services at syringe exchange program
Groups:
- Health Education Plus Incentives for Abstinence: Participants in the health education plus incentives for abstinence condition will have the opportunity to earn financial incentives for abstaining from stimulant use. Additionally, they also receive the health education provided in the Health Education condition, with sessions consisting of an educational program addressing a variety of health, wellness, and lifestyle topics adapted from a previously implemented wellness manual.
Period: Overall Study
Arm/Group | Health Education | Health Education Plus Incentives for Abstinence
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Education | Health Education Plus Incentives for Abstinence | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 6 | 10 | 16
  Sex/Gender: Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 11 | 12 | 23
  Race/Ethnicity: Latinx/Hispanic & Black & American Indian/Alaska Native | 0 | 1 | 1
  Race/Ethnicity: White & American Indian/Alaska Native | 1 | 1 | 2
  Race/Ethnicity: White & Black/African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stimulant Free Urine Sample
Description: all samples will be assessed using point-of-care test urine drug test conducted at the center
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: % stimulant-negative urine drug test
Units Other Than Participants: Urine drug test
Arm/Group | Health Education | Health Education Plus Incentives for Abstinence
Number analyzed (Participants) | 13 | 14
Number analyzed (Urine drug test) | 312 | 336
% stimulant-negative urine drug test | 6.1 (2.7) | 23.6 (10.3)

ADVERSE EVENTS:
Time Frame: From enrollment to study completion at 12 weeks
Arm/Group | Health Education | Health Education Plus Incentives for Abstinence
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
This project was designed as a pilot study with a small sample size. As such, there are limitations of the statistical power due to the small sample size. Although the originally proposed sample size by condition was not met, the results are able to discern patterns of differences in the primary outcome by study condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT05787847/Prot_SAP_000.pdf